CLINICAL TRIAL: NCT01449175
Title: A Registry Study of the AeriSeal® System or Lung Volume Reduction in Patients With Advanced Emphysema
Status: Terminated | Type: Observational
Sponsor: Aeris Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: 03-C11-001PLV
Record Dates: First submitted 2011-04-19; First posted 2011-10-10 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Pulmonary Obstructive Disease; Emphysema
Keywords: AeriSeal; treatment; device; breathing; COPD; emphysema; polymeric lung volume reduction (PLVR); biologic lung volume reduction (BLVR); heterogeneous; homogeneous; Respiratory Tract Diseases; Lung Diseases; Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Respiratory Aspiration; Respiratory Tract Diseases; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to provide post market clinical follow-up (PMCF) to obtain long term safety and efficacy information about the AeriSeal System treatment in patients with advanced emphysema.

DETAILED DESCRIPTION:
The purpose of this study is to provide post market clinical follow-up (PMCF) to obtain long term safety and efficacy information about the AeriSeal System treatment in patients with advanced homogeneous or heterogeneous emphysema.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of completion of Aeris' post market follow-up Continuation Study, 03-C10-001PLV.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients participating in the Registry Study must have been enrolled in either Group 4 (homogeneous emphysema) or Group 5 (heterogeneous emphysema) of Aeris' Investigational Study 03-C08-003PLV and completed 48 week follow-up in the AeriSeal post market follow-up Continuation Study (03-C10-001PLV).
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in number of Serious Adverse Events (SAE) | Weeks 48, 96, 120, 144 following treatment
  Count number of SAEs during weeks: 48, 96, 120, 144 as a function of long term safety

SECONDARY OUTCOMES:
Change in Vital Signs | weeks 48, 96, 120, 144 following treatment
  Change from baseline at 48, 96, 120 and 144 weeks of Vital Signs
Change in Oxygen (O2) Use | Weeks 48, 96, 120, 144 following treatment
  Change in amount of O2 used (at rest, with activity, during sleep) in weeks 48, 96, 120 and 144 from baseline.
Change in medications | week 48, 96, 120, 144 following treatment
  Change in medication regiment in weeks 48, 96, 120 and 144 from baseline.
Change in Pulmonary Function Tests (PFT) | Weeks 48, 96, 120, 144 following treatment
  Change in PFT (Spirometry, Diffusing Capacity, Plethysmograpy) in weeks 48, 96, 120 and 144 from baseline
Change in notable radiology results | weeks 48, 96, 120, 144 following treatment
  Change in notable radiology results (infiltrates, mass lesions, pleural abnormalities) from baseline in weeks 48, 96, 120 and 144.

CONTACTS AND LOCATIONS:
Locations (8):
- Otto Wagner Spital Wien, Wein, Austria
- Service de Pneumologie, Hôpital Pasteur, Centre Hospitalier Universitaire de Nice, Nice, France
- Germany (4):
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Thoraxklinik Heidelberg, Heidelberg
  - LungenKlinik Hemer, Hemer
  - LMU Medizinische Klinik und Poliklinik Klinikum Großhadern, München
- Israel (2):
  - Soroka Medical Center, Beer Sheeva
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva